CLINICAL TRIAL: NCT03718091
Title: A Phase II Study of M6620 (VX-970) in Selected Solid Tumors
Brief Title: M6620 (VX-970) in Selected Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Gregory Cote, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-274
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor; Leiomyosarcoma; Osteosarcoma
Keywords: Solid Tumor; leiomyosarcoma; Osteosarcoma
MeSH Terms: conditions — Leiomyosarcoma; Osteosarcoma | interventions — berzosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort T1: ATRX-mutant Leiomyosarcoma (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort T2: Truncating ATM Mutation (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort T3: Other HR Gene Mutations (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 1A: Osteosarcoma (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 1B: Leiomyosarcoma (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 2: Truncating ATM mutation (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 3A: Germline BRCA mutation (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 3B: Other HR Alteration (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 4A: MYC amplification, FBXW7 mutation (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 4B: Cyclin E amplification (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort 5: ARID1A mutation (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620
- Cohort T4: SDH-Mutant GIST (Experimental): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  Interventions: Drug: M6620

INTERVENTIONS:
Drug: M6620 — M6620 is a drug designed to inhibit the ATR enzyme. Inhibiting ATR may block how cancers repair their naturally damaged DNA, handle cancer cell stress, and maintain cancer cell life and health.
  Other Names: VX-970

SUMMARY:
This research study is studying a drug called M6620 as a possible treatment for advanced solid tumor.

DETAILED DESCRIPTION:
This study is made up of two phases: a Translational Lead-In Phase and a Phase II. These two phases serve different functions. The translational lead-in phase is designed to test the drug on a small number of patients in efforts to gain information on two research questions:

* If M6620 has an anti-cancer effect on participants
* If M6620 research findings that were discovered in laboratory studies are also found in human research studies.

Phase II is a much larger study to determine if M6620 has an anti-cancer effect in different groups of patients.

The FDA (the U.S. Food and Drug Administration) has not approved M6620 as a treatment for any disease.

ATR is an enzyme in cells that is responsible for multiple functions including repairing damaged DNA, helping cells that are stressed during the DNA copying process, and working to maintain the ends of chromosomes. In cancer cells, active ATR enzymes protect the cancer by helping the cells repair damage, stay alive, and maintain health. M6620 is a drug designed to inhibit the ATR enzyme. Inhibiting ATR may block how cancers repair their naturally damaged DNA, handle cancer cell stress, and maintain cancer cell life and health. Administration of M6620 may therefore assist in the slowing of growth or destruction of some cancers.

In this research study, the investigators are...

* Gathering initial data on the anti-cancer activity of M6620 when given alone to participants within selected cancer populations
* Determining if there are changes in the biological components in the participant's body that may be associated with damaged DNA repair

ELIGIBILITY:
Inclusion Criteria:

Participants Enrolling to the Translational Lead-in Study:

* For enrollment to cohort T1: participants must have metastatic or progressive LMS with a) treatment with at least one prior systemic therapy b) ATRX mutation by NGS
* For enrollment to cohorts T2 or T3: participants must have a histologically or cytologically confirmed advanced solid tumor for which no standard curative therapy is available.
* For enrollment to cohort T2: participants must have a truncating ATM mutation. Testing may be completed via the DFCI/BWH OncoPanel, MGH SNaPshot, or any other CLIA-certified method.
* For enrollment to cohort T3, participants must have one of the following (testing may be completed via the DFCI/BWH OncoPanel, MGH SNaPshot, or any CLIA-certified laboratory):

  * Germline mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function).
  * A somatic mutation in BRCA1 or BRCA2, or another mutation within a known HR gene including BARD1, BRIP1, CDK12, CHEK2, FANCA, FANCC, FANCE, FANCF, FANCM, MRE11A, NBN, PALB2, RAD51B, RAD51C, or RAD51D.
  * A MYC amplification of greater than 6-fold.
  * FBXW7 truncating or missense mutation designated as deleterious.
  * CCNE1 amplification of greater than 8-fold.
  * An ARID1A mutation as determined by the DFCI/BWH OncoPanel or any other CLIA-certified method.
  * Other (unlisted) mutations within known HR genes may be considered with approval from the site principal investigator.
* For enrollment to cohort T4: participants must have GIST with known mutation in SDHX genes or loss of expression of SDHX protein(s), as determined by standard pathology assays. Prior therapy is not required.
* Age ≥ 18 years
* ECOG performance status ≤ 2 (Karnofsky [KPS] ≥ 60%; KPS of 50 is not permitted)
* Participants must have tumor amenable to biopsy, and be a candidate for tumor biopsy according to the treating investigator. The patient must be willing to undergo a fresh tumor biopsy for this study.
* Participants must have archival tissue available for analysis. Participants without available archival tissue enrolling to the translational lead-in study may instead use tissue from the fresh pre-treatment biopsy.

Participants Enrolling to the Phase II:

* For enrollment to cohort 1A: participants must have metastatic or progressive osteosarcoma treated with at least one prior systemic therapy.
* For enrollment to cohort 1B: participants must have metastatic or progressive leiomyosarcoma treated with at least one prior systemic therapy.
* For enrollment to cohorts 2 - 5: participants must have a histologically or cytologically confirmed advanced solid tumor for which no standard curative therapy is available.
* For enrollment to cohort 2: participants must have a truncating ATM mutation. Testing may be completed via the DFCI/BWH OncoPanel, MGH SNaPshot, or any other CLIA-certified method.
* For enrollment to cohort 3A: participants must have a germline mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function). Testing may be completed via the DFCI/BWH OncoPanel, MGH SNaPshot, or any CLIA-certified laboratory.
* For enrollment to cohort 3B: participants must have a somatic mutation in BRCA1 or BRCA2, or another mutation within a known HR gene including BARD1, BRIP1, CDK12, CHEK2, FANCA, FANCC, FANCE, FANCF, FANCM, MRE11A, NBN, PALB2, RAD51B, RAD51C, or RAD51D. Other (unlisted) mutations within known HR genes may be considered with approval from the site principal investigator.
* For enrollment to cohort 4A: participants must have a MYC amplification of greater than 6-fold or an FBXW7 truncating or missense mutation designated as deleterious, as determined by the DFCI/BWH OncoPanel, MGH SNaPshot, or any other CLIA-certified method.
* For enrollment to cohort 4B: participants must have a CCNE1 amplification of greater than 8-fold as determined by the DFCI/BWH OncoPanel, MGH SNaPshot, or any other CLIA-certified method.
* For enrollment to cohort 5: participants must have an ARID1A mutation as determined by the DFCI/BWH OncoPanel, MGH SNaPshot, or any other CLIA-certified method.
* For enrollment to cohort 1A: Age > 12
* For enrollment to cohorts 1B - 5: Age ≥ 18
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%; KPS of 50 is not permitted) for participants ≥ 16 years of age, Lansky ≥ 50% for participants < 16 years of age
* Participants must have archival tissue available for analysis

All Participants:

* If any participant could enroll to more than one cohort based on mutational status, the cohort enrollment decision will be discussed with the overall principal investigator. For example, if a participant has both an ATM mutation and an FBXW7 mutation and thus could enroll to either Cohort 2 or Cohort 4A, the decision of which cohort to enroll to will be made in conjunction with the overall principal investigator. The decision as to which cohort the participant should be enrolled on must be made prior to the initiation of study treatment.
* Participants must have RECIST 1.1 measurable disease.
* Participants must have normal organ and marrow function as defined below:

All Participants:

* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) for age

Adult Participants (Age ≥ 18 years):

* AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN; OR

  * 5 × institutional ULN if liver metastases are present
* Serum or plasma creatinine ≤ 1.5 × institutional ULN, OR
* Creatinine clearance ≥ 60 mL/min by Cockcroft-Gault equation for participants with creatinine levels above 1.5 × institutional ULN

Pediatric Participants (Age < 18 years):

* ALT (SGPT) ≤ 3 × institutional (ULN)

  -for the purposes of this study, the ULN for SGPT will be defined as 45 U/L.
* Serum or plasma creatinine Participants 13 - 15 years: males ≤ 1.5 mg/dL, females

  ≤ 1.4 mg/dL, participants 16 - 17 years: males ≤ 1.7 mg/dL, females ≤ 1.4 mg/dL; OR
* Creatinine clearance ≥ 60 mL/min/1.73 m2 by Schwartz formula for participants with creatinine levels above the limits described above

  * The effects of M6620 on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of M6620 administration.
  * Ability to understand and the willingness to sign a written informed consent document (or parent or legally authorized representative, if minor).

Exclusion Criteria:

* Participants who have had chemotherapy, immune therapy, other investigational therapy, major surgery, or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or participants who have not recovered to ≤ Grade 1 or baseline from therapies administered more than 3 weeks prior (with the exceptions of 1. Alopecia and peripheral neuropathies which may be ≤ Grade 2 at study entry and 2. Laboratory abnormalities that are not listed in 3.1 and that are not considered clinically meaningful [e.g. decreased lymphocyte count, electrolyte abnormalities]
* Participants who have received oral tyrosine kinase inhibitors (TKIs) within 5 half-lives of study entry.
* Participants who have previously received treatment with an ATR inhibitor, including but not limited to M6620 (VX-970).
* Participants with known untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with a history of brain metastases that have been treated, no longer require corticosteroids, and have been stable on imaging for at least one month following the end of treatment are permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because M6620 is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620, breastfeeding should be discontinued if the mother is treated with M6620.
* Known HIV-positive participants are ineligible because of the increased risk of lethal infections when treated with potentially marrow-suppressive therapy.
* Patients with a history of another malignancy are excluded with the exception of 1. patients who remain disease-free for 3 years and 2. adequately treated cervical carcinoma in situ, non-melanoma skin cancer (e.g. basal cell, squamous cell carcinomas), low-risk thyroid cancer.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Cote, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Children Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original study was a planned molecular lead-in followed by a basket study (6 per cohort x4 cohorts; 24 total). 6 patients were replaced as they either did not receive study drug or were unable to complete paired biopsies (replacement permitted per protocol). Thus, Cohorts T1,T2, and T3 have >6 pts. One patient slot was not accrued for T4.
  The basket study was not opened due to lack of efficacy in the lead-in.
Groups:
- Cohort T3: Other HR Gene Mutations and Replicative Stress; Cohort T4: SDH-Mutant GIST: M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  M6620: M6620 is a drug designed to inhibit the ATR enzyme. Inhibiting ATR may block how cancers repair their naturally damaged DNA, handle cancer cell stress, and maintain cancer cell life and health.
Period: Overall Study
Arm/Group | Cohort T1: ATRX-mutant Leiomyosarcoma | Cohort T2: Truncating ATM Mutation | Cohort T3: Other HR Gene Mutations and Replicative Stress | Cohort T4: SDH-Mutant GIST
Started | 8 | 7 | 9 | 5
Completed | 8 | 7 | 9 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort T1: ATRX-mutant Leiomyosarcoma | Cohort T2: Truncating ATM Mutation | Cohort T3: Other HR Gene Mutations and Replicative Stress | Cohort T4: SDH-Mutant GIST | Total
Number analyzed (Participants) | 8 | 7 | 9 | 5 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 4 | 4 | 18
  >=65 years | 2 | 3 | 5 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 3 | 1 | 16
  Male | 0 | 3 | 6 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 7 | 6 | 4 | 24
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 6 | 9 | 3 | 25
  More than one race | 1 | 1 | 0 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Phospho-Chk1 Levels in Biopsy Specimens
Description: Changes in the levels of Phospho-Chk1 in biopsy specimens of patients treated with M6620 monotherapy from baseline to cycle 1 day 15. This is a pharmacodynamic endpoint to evaluate target engagement. Results are in percent change of Phospho-Chk1 levels from baseline versus on-treatment biopsies.
Time Frame: Baseline, Day 15
Population: change in phospho-Chk1
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort T1: ATRX-mutant Leiomyosarcoma | Cohort T2: Truncating ATM Mutation | Cohort T3: Other HR Gene Mutations | Cohort T4: SDH-Mutant GIST
Number analyzed (Participants) | 5 | 3 | 4 | 1
percent change | 156 [-45 to 511] | 196 [131 to 272] | 89 [-36 to 603] | 84 [84 to 84]

2. Primary Outcome: Change in yH2AX Levels in Biopsy Specimens
Description: Changes in the levels of yH2AX in biopsy specimens of patients treated with M6620 monotherapy from baseline to cycle 1 day 15.
Time Frame: Baseline, Day 15
Population: paired biopsies
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort T1: ATRX-mutant Leiomyosarcoma | Cohort T2: Truncating ATM Mutation | Cohort T3: Other HR Gene Mutations | Cohort T4: SDH-Mutant GIST
Number analyzed (Participants) | 5 | 3 | 4 | 1
percent change | -36.8 [-83.9 to 820.4] | 142.2 [-40.5 to 395.9] | -34.3 [-50.9 to 114.5] | -30.8 [-30.8 to -30.8]

3. Primary Outcome: Disease Control Rate
Description: The number of participants that achieve either Stable Disease (SD), Partial Response (PR), or Complete Response (CR) at 16 weeks.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 16 weeks
Measure: Number; unit: absolute # pts with CR/PR/SD at 16 wks
Arm/Group | Cohort T1: ATRX-mutant Leiomyosarcoma | Cohort T2: Truncating ATM Mutation | Cohort T3: Other HR Gene Mutations | Cohort T4: SDH-Mutant GIST
Number analyzed (Participants) | 8 | 7 | 9 | 5
absolute # pts with CR/PR/SD at 16 wks | 0 | 0 | 0 | 2

4. Secondary Outcome: Number of Participants With Treatment Related Serious Adverse Events
Description: Adverse events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE 5.0)
Time Frame: AE data was collected from cycle 1 day 1 until 30 days after last dose or resolution of the AE.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort T1-T4 (Analyzed Together for AEs): M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  M6620: M6620 is a drug designed to inhibit the ATR enzyme. Inhibiting ATR may block how cancers repair their naturally damaged DNA, handle cancer cell stress, and maintain cancer cell life and health.
  AEs were analyzed in aggregate. There is are no data suggesting that the AE profile would be different between tumor molecular lesion in this heterogeneous population.
Arm/Group | Cohort T1-T4 (Analyzed Together for AEs)
Number analyzed (Participants) | 29
Participants | 12

ADVERSE EVENTS:
Time Frame: AE data was collected from cycle 1 day 1 until 30 days after last dose or resolution of the AE. The study length for collection of AEs was 575 days total.
Description: An AE is any untoward medical occurrence in a patient or clinical study subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  AE analyzed together in this heterogeneous population.
Groups:
- Cohorts T1-4: M6620 will administered intravenously on days 1,4, 8, 11, 15, 18, 22, 25 on a 28-day cycle.
  M6620: M6620 is a drug designed to inhibit the ATR enzyme. Inhibiting ATR may block how cancers repair their naturally damaged DNA, handle cancer cell stress, and maintain cancer cell life and health.
Arm/Group | Cohorts T1-4
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 12/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts T1-4 (N=29)
grade 4 elevated AST (Hepatobiliary disorders) | 1 (1) — elevated AST
grade 3 AST increase (Hepatobiliary disorders) | 2 (2)
grade 2 alkaline phosphatase increase (Hepatobiliary disorders) | 2 (2)
elevated bilirubin (Hepatobiliary disorders) | 1 (1)
grade 3 anemia (Blood and lymphatic system disorders) | 1 (1)
grade 3 anaphylaxis (Immune system disorders) | 1 (1)
grade 3 febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
grade 3 ALT increase (Hepatobiliary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03718091/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03718091/ICF_001.pdf